CLINICAL TRIAL: NCT06771167
Title: NYC Community Engagement Alliance (NYCEAL) Against COVID-19 Disparities
Brief Title: Building Community Resilience Program
Acronym: BCR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Carol R Horowitz, Dean for Gender Equity in Science and Medicine, Professor of Population Health Science and Policy, Professor of Medicine, General Internal Medicine, Icahn School of Medicine at Mount Sinai
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GCO 21-0396; HL158287 (Other Grant/Funding Number: NYU's MPI NIH CEAL)
Record Dates: First submitted 2025-01-07; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Resilience, Psychological; Burnout, Psychological; Stress, Psychological
Keywords: Resilience; Community Health Workers; Burnout; Emotional Well-Being; Educational Workshops; Community-Based Organizations
MeSH Terms: conditions — Burnout, Psychological; Stress, Psychological

STUDY DESIGN:
Intervention Model Description: The researchers will employ a quasi-experimental pre-post non-equivalent waitlist control group design to proactively minimize logistical barriers, maximize feasibility of implementing the intervention, and reduce ethical concerns of depriving communities of beneficial interventions. The waitlist control sites (the second cohort of CBOs receiving the educational workshops) are expected to have similar sociodemographic characteristics and health burdens as the intervention sites. Data collection in the second cohort of sites will allow the researchers to examine whether observed changes in outcomes are attributable to the intervention and ensure that all of the partnering CBO sites have access to BCR educational workshops for CHWs and frontline workers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate Intervention Group (First Cohort) (Experimental): The first cohort of up to 36 participants will complete two surveys: a baseline survey within one month before the workshops begin, and a post-test survey within one month after the final workshop (approximately 8 months total from first to last survey)
  Interventions: Behavioral: Building Community Resilience Program (BCR)
- Waitlist Group (Second Cohort) (Experimental): The second cohort of up to 36 participants will complete four surveys: two surveys in year 1 (matching the timing of the first cohort's surveys to serve as a control group), and two additional surveys in year 2 when they receive the intervention (a baseline survey within one month before their workshops begin, and a post-test survey within one month after their final workshop).
  Interventions: Behavioral: Building Community Resilience Program (BCR)

INTERVENTIONS:
Behavioral: Building Community Resilience Program (BCR) — To improve CHW resilience and wellbeing, during each BCR cycle, the 6 participating CBOs will send groups of four to six CHWs to six virtual, hour-long, evidence-based interactive workshops (48-72 CHWs over the 2 cycles).

SUMMARY:
Established in 2021, NYCEAL consists of approximately 40 organizational partners and 120 Community Health Workers (CHWs). Over the next four years (2024-2028), NYCEAL will work with this network to implement the following intervention: Building Community Resilience Program (BCR). To assess the impact of this intervention, an implementation research framework will be used, and pre- and post-surveys conducted, and other process evaluation measures collected. Changes in outcomes measures such as stress, resilience, overall wellbeing, and other related outcomes for participants in the BCR program will be measured for community healthcare workers and/or frontline workers that receive educational workshops.

DETAILED DESCRIPTION:
BCR Study Design and Methods: To incorporate adequacy and plausibility, approaches in public health research often move beyond randomized trials to better support evaluation and public health decision-making, while being responsive to the three hallmarks of sound study design: minimizing selection and information bias, controlling confounding, and ruling out chance. BCR will leverage a quasi-experimental approach to evaluate the impact of the proposed intervention on participating NYCEAL CBOs' CHWs. The researchers will employ a pre-post non-equivalent waitlist control group design to proactively minimize logistical barriers, maximize feasibility of implementing the intervention, and reduce ethical concerns of depriving communities of beneficial interventions. The waitlist control sites (the second cohort of CBOs receiving the educational workshops) are expected to have similar sociodemographic characteristics and health burdens as the intervention sites. Data collection in the second cohort of sites will allow the researchers to examine whether observed changes in outcomes are attributable to the intervention and ensure that all of the partnering CBO sites have access to BCR educational workshops for CHWs and frontline workers. The researchers will assess impact using an outcomes survey co-developed with NYCEAL CBO partners (not individuals receiving the intervention). The researchers will conduct surveys via RedCap at pre- and 6-month post-intervention timepoints with CHWs at BCR sites (for both cohorts). The primary outcome for the CHW intervention is burnout (Mini-Z burnout scale), which is closely linked to workforce retention, work quality, and client interactions. Secondary outcomes include validated measures for resilience, stress, worker wellbeing, and job satisfaction. BCR intervention sites were chosen based on interest, history of collaboration, readiness, capacity and interest in promoting resilience, and consequently overall good health at the organizational level, and as they serve priority populations in high disparity neighborhoods (and the wellbeing of these sites is important for continuing the work of supporting local communities).

The BCR educational workshops will take place over two years, with two cohorts of six CBOs each (12 CBOs total). Both cohorts will be recruited simultaneously, with the second cohort serving as a waitlist control group during the first year. To improve CHW resilience and wellbeing, during each BCR cycle, the 6 participating CBOs will send groups of four to six CHWs to participate in the program (48-72 CHWs over the 2 cycles). Each cohort will receive six virtual, hour-long, evidence-based interactive workshops, delivered once per month over a six-month period. The first cohort will receive the intervention in year 1, while the second cohort will receive the intervention in year 2.

Topics include: 1) realistic optimism ("Build Your Hope"); 2) active coping and facing fears ("Face Your Fears"); 3) self-care ("Mind Your Body"); 4) social support and networks ("Mind Your Circle"); 5) building our "why" ("Mind Your Purpose"); and 6) addressing social justice ("Mind Your Community"). DePierro and an experienced social worker will co-facilitate the interactive, skills based workshops. They will include information in lay format about the importance of resilience factors and activities that result in the development of resilience plans. For example, activities to support the development of "utilizing social support networks"include building/mapping a social support network tree that allows people to take stock of the areas of support needed to further cultivate, and develop action-oriented SMART goals that address specific needs. Workshop participants will also have free access to a mobile app (Wellness Hub) that was developed by DePierro they can use to reinforce these topics through maintenance activities.

ELIGIBILITY:
Inclusion Criteria:

* Able to consent
* Able to fill out the screening RedCap short survey
* Have access to a computer or smart gadget that will allow participant to be able to join the zoom call
* English speaking
* Living in NYC (5 boroughs)
* 18+ years of age (no upper bound age limit)
* Working with an NYCEAL CBO participating in BCR programming

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Incapacitated to an extent that they are unable to comprehend a conversation or communicate effectively in a group setting
* Unable to consent to be part of the study
* Does not have access to a computer or smart gadget that will allow participant to be able to join the zoom call
* Does not speak English
* Not living in NYC
* Not 18+ years of age
* Not working with an NYCEAL CBO participating in BCR programming

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Mini-Z Burnout Scale Score | Baseline (within one month before workshops begin) and post-test (within one month after workshops end at 6 months)
  The Mini Z Burnout Inventory score measures burnout and is calculated by summing responses from all 10 questions, with possible scores ranging from 10 to 50. Higher scores indicate a more positive and joyful work environment, with scores of 40 or above representing a joyful workplace.

SECONDARY OUTCOMES:
The Mount Sinai Resilience Scale Scores | Baseline (within one month before workshops begin) and post-test (within one month after workshops end at 6 months)
  The Mount Sinai Resilience Scale (MSRS) measures resilience with scores ranging from 0 to 144. Scores of 45 or higher may indicate average or above-average resilience levels. Higher scores indicate higher level of resilience.
NIOSH Worker Well-being Questionnaire - Stress | Baseline (within one month before workshops begin) and post-test (within one month after workshops end at 6 months)
  The stress measure consists of 4 selected items from the NIOSH Worker Well-being Questionnaire (WellBQ). The overall stress score is calculated as the average of these 4 items, with scores above the midpoint indicating high stress levels. Responses are indicated on a 7-item Likert scale from. Full scale from 1-7. Higher scores indicate stronger feelings of collegial support.
NIOSH Worker Well-being Questionnaire - Collegial Support | Baseline (within one month before workshops begin) and post-test (within one month after workshops end at 6 months)
  Collegial Support is measured using 9 items from the NIOSH Worker Well-being Questionnaire (WellBQ). Responses are indicated on a 5 point Likert scale with '1' being "Strongly Disagree", '4' being "Strongly Agree", and '5' being "Does not apply". Full scale from 1-5. Higher scores indicate stronger feelings of collegial support.
NIOSH Worker Well-being Questionnaire - Meaningful Work | Baseline (within one month before workshops begin) and post-test (within one month after workshops end at 6 months)
  Meaningful work is measured using 2 selected items from the NIOSH Worker Well-being Questionnaire (WellBQ). Responses are indicated on a 5 point Likert scale with '1' being "Strongly Disagree", '4' being "Strongly Agree", and '5' being "Does not apply". Full scale from 1-4. Higher scores indicate stronger feelings of engaging in meaningful work.
NIOSH Worker Well-being Questionnaire - Fair/Equitable Compensation | Baseline (within one month before workshops begin) and post-test (within one month after workshops end at 6 months)
  Fair/equitable job compensation is measured using 1 selected items from the NIOSH Worker Well-being Questionnaire (WellBQ). The response is indicated on a 5 point Likert scale with '1' being "Strongly Disagree", '4' being "Strongly Agree", and '5' being "Does not apply". Higher scores indicate stronger feelings of fair compensation.
NIOSH Worker Well-being Questionnaire - Job Security | Baseline (within one month before workshops begin) and post-test (within one month after workshops end at 6 months)
  Job security is measured using 1 selected items from the NIOSH Worker Well-being Questionnaire (WellBQ). The response is indicated on a 5 point Likert scale with '1' being "Strongly Disagree", '4' being "Strongly Agree", and '5' being "Does not apply". Higher scores indicate stronger feelings of job security.

CONTACTS AND LOCATIONS:
Overall Officials: Carol Horowitz, MD, MPH, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
The researchers will not be sharing IPD, all results will be in aggregate.